CLINICAL TRIAL: NCT06368375
Title: Clinical and Genetic Findings in Patients With PRPF31-associated Retinitis Pigmentosa
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: PRPF31-3102022BO2
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; PRPF31; inherited retinal dystrophy; carrier
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective chart review study to elucidate the genotype and phenotype of patients with PRPF31-associated retinitis pigmentosa and asymptomatic carriers of the respective variant(s)

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed PRPF31-associated inherited retinal dystrophy or asymptomatic carrier of the respective variant(s)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with genetically confirmed PRPF31-associated inherited retinal dystrophy or asymptomatic carrier of the respective variant(s)
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | September 2007 - January 2022
  best corrected visual acuity
Visual Field (VF) | September 2007 - January 2022
  visual field as measured by semi-automated 90° kinetic visual field exam using target III4e
Fundus Photography (FP) | September 2007 - January 2022
  characterization of the retina with fundus photography
Optos | September 2007 - January 2022
  characterization of the retina with ultra-wide-field scanning laser ophthalmoscopy
Autofluorescence (AF) | September 2007 - January 2022
  characterization of the retina with fundus autofluorescence
Optical Coherence Tomography (OCT) | September 2007 - January 2022
  characterization of the retina with optical coherence tomography, e.g. foveal ellipsoid zone loss
Full-Field Electroretinogram (ff-ERG) | September 2007 - January 2022
  characterization of retinal function with full-field electroretinogram

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kuehlewein, MD, Principal Investigator — Department for Ophthalmology, University of Tuebingen; Susanne Kohl, PhD, Principal Investigator — Molecular Genetics Laboratory, Department for Ophthalmology, University of Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No